CLINICAL TRIAL: NCT05879575
Title: Effects and Pathophysiology of Weight Training on Pregnancy-related Pelvic Girdle Pain (PPGP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Collaborators: National Taiwan University Hospital (Other); National Taiwan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111-152-F
Record Dates: First submitted 2023-03-01; First posted 2023-05-30 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Pelvic Girdle Pain
Keywords: pregnancy-related pelvic girdle pain; weight training; resistance training
MeSH Terms: conditions — Pelvic Girdle Pain | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: intervention group: receive weigh training during 16-36 gestational weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): receive weight training during 16-36 gestational weeks and observe pain condition
  Interventions: Behavioral: weight training
- control group (No Intervention): observe pain condition

INTERVENTIONS:
Behavioral: weight training — Pregnant women assigned to the intervention group will receive online weight training sessions twice a week, for 60 minutes per session, from the 16th to the 36th week of pregnancy. The Pelvic Girdle Questionnaire will be used to assess the condition of pelvic girdle pain during pregnancy, and to analyze whether weight training can improve this problem. Pelvic floor muscle structure will also be analyzed by pelvic ultrasound to determine whether it has been altered by weight training, leading to an improvement in pain.
  Arms: intervention group

SUMMARY:
In recent years, due to the popularity of exercise during pregnancy, the American College of Obstetricians and Gynecologists recommends that pregnant women should engage in 150 minutes of moderate-intensity exercise per week, including aerobic exercise or weight training. This can help reduce pregnancy complications (such as preeclampsia, gestational diabetes, pelvic pain, etc.) and does not increase the risk of miscarriage or premature birth. Pelvic pain during pregnancy is the most troublesome problem for pregnant women, often affecting their daily lives and mental health, leading to the need for long-term use of painkillers and even affecting their daily routine and sleep. Currently, research has also found that exercise during pregnancy can improve pelvic pain during pregnancy and reduce the inconvenience caused by pain in daily life. However, weight training can strengthen spinal stability and reduce lower back pain problems in non-pregnant individuals, but there is currently no research discussing whether weight training for pregnant women can improve pelvic pain during pregnancy, possibly because weight training for pregnant women is not widely accepted by society and is often associated with misconceptions and prejudices. Recent literature synthesis analysis tells us that weight training during pregnancy does not increase the risk of premature birth or miscarriage. Pregnant women in supervised moderate-intensity weight training do not endanger the health of the mother or fetus, and the safety is sufficient. Therefore, we hope to understand the effects and mechanisms of weight training during pregnancy on pelvic pain during pregnancy through this study.

DETAILED DESCRIPTION:
Pregnancy-related pelvic girdle pain is one of the most troubling issues for pregnant women. Everyday activities, such as walking, standing, sitting, and even lying down, can potentially trigger or exacerbate the pain. The diagnostic criteria for pelvic girdle pain are relatively complex. Since the 2008 European guidelines suggested clinical physiotherapy test conditions, they have gradually been adapted for pregnant women. In 2021, Monika revised the diagnostic criteria, allowing pregnant women to self-check for pelvic girdle pain diagnosis, with the following self-test conditions:

Pregnant women have experienced at least one day in the past four weeks when pelvic girdle pain has affected their daily lives.

They can clearly point out the painful area (e.g., sacroiliac joint or pubic symphysis joint pain).

At least one positive anterior pelvic girdle pain test item, or two positive posterior pelvic girdle pain test items, are confirmed through a "pelvic girdle pain self-check." Research has found that 50-70% of pregnant women experience pelvic girdle pain during pregnancy, with 33%-50% experiencing pain even before 20 weeks of gestation. However, 7% continue to have pelvic girdle pain issues for life after childbirth. Pregnancy-related pelvic girdle pain affects daily life and mental health, often leading to long-term use of painkillers and affecting daily routines and sleep.

Recent research suggests that weight training can strengthen spinal stability and reduce lower back pain in non-pregnant individuals. The American College of Obstetricians and Gynecologists recommends pregnant women engage in 150 minutes of moderate-intensity exercise per week, including aerobic exercise or weight training. Studies also show that exercising during pregnancy can improve pelvic girdle pain, reducing inconvenience in daily life, but it cannot reduce the incidence of pain.

In a 2019 survey about pregnancy-related pain, 47% of pregnant women reported having lower back pain during pregnancy. The study found that the fewer times women exercised per week before pregnancy, the more likely they were to experience lower back pain during pregnancy.

However, most current exercise intervention studies for pregnancy-related pelvic girdle pain focus on aerobic exercise rather than weight training. Weight training for pregnant women has not yet been widely accepted, and there are many misconceptions. However, meta-analysis of literature shows that weight training during pregnancy does not increase the risk of preterm birth or miscarriage. Moderate-intensity weight training under guidance does not harm maternal or fetal health, and its safety is sufficient. Therefore, we want to understand whether weight training, as opposed to traditional aerobic exercises, can improve pregnancy-related pelvic girdle pain. Are there differences in muscle cell proliferation and differentiation during pregnancy compared to non-pregnant adults? Does incomplete muscle cell differentiation affect muscle strength, leading to pain in pregnant women? And what mechanisms do weight training exercises use to improve pain?

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are within 14 weeks of gestation and carrying a single fetus.
* Pregnant women who can clearly identify the location of their pelvic girdle pain (e.g. sacroiliac joint or pubic symphysis pain).
* Pregnant women who have at least one positive result in a front pelvic girdle pain test or two positive results in a back pelvic girdle pain test based on the "Self-Administered Pelvic Girdle Pain Test".
* Pregnant women assigned to the intervention group must be able to comply with the exercise program.
* Pregnant women assigned to the control group must not engage in weight training.

Definition of weight training: The use of resistance to induce muscular contraction, with the goal of increasing strength and endurance of the muscles. This can be achieved systematically using weights, such as one's own body weight, or equipment that provides resistance to muscle contraction, such as dumbbells, barbells, or resistance bands.

- Participants will receive follow-up care and delivery at National Taiwan University Hospital in Hsinchu.

Exclusion Criteria:

* For pregnant women with twins or multiple pregnancies
* With any pregnancy exercise contraindications from the American College of Obstetricians and Gynecologists, including:

  * Pre-existing internal medical conditions such as severe unstable heart disease, restrictive lung disease, symptomatic severe anemia, poorly controlled hypertension, poorly controlled diabetes, poorly controlled thyroid disease, and other similar conditions.
  * Pregnancy-related conditions such as early rupture of membranes, signs of preterm labor, incomplete cervix closure, history of cervical cerclage, habitual miscarriage, and previous history of preterm birth.
* History of spinal or pelvic surgery
* Known pelvic pain before pregnancy, such as lumbar or pelvic fractures or chronic pain caused by previous surgery
* Clear diagnosis of pre-pregnancy back pain causes, such as herniated discs or nerve root diseases
* Regular use of pain relief medications before pregnancy, such as acetaminophen, non-steroidal anti-inflammatory drugs (NSAIDs), morphine, and platelet-rich plasma (PRP) therapy
* Regular weight training habit before enrollment (at least twice a week)
* Not planning to give birth at National Taiwan University Hospital
* Already participating in other interventional clinical trials.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 70 (Estimated)
Dates: Start 2023-05-31 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
PGQ score | change of the PGQ score between the first trimester (before GA 14 weeks) and the third trimester before delivery (GA 35 to 36+6 weeks)
  The main evaluation indicators will include the PGQ activity assessment to evaluate the impact of pelvic girdle pain on daily life, and the PGQ symptom assessment to evaluate the severity of symptoms. These indicators will be used to assess whether weight training during pregnancy improves pelvic girdle pain.

SECONDARY OUTCOMES:
Cervical length | difference of the cervical length between the first trimester (before GA 14 weeks) and the third trimester (GA 35 to 36+6 weeks) of the pregnancy
  To evaluate whether exercise during pregnancy may shorten the cervical length.
Duration of the first stage of labor | During labor
  To evaluate whether exercise during pregnancy may effect the duration of the first stage of labor
Duration of the second stage of labor | During labor
  To evaluate whether exercise during pregnancy may effect the duration of the second stage of labor

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Yuan Li, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Physical Activity and Exercise During Pregnancy and the Postpartum Period: ACOG Committee Opinion, Number 804. Obstet Gynecol. 2020 Apr;135(4):e178-e188. doi: 10.1097/AOG.0000000000003772. PMID 32217980
- [Background] Bentzinger CF, Wang YX, Rudnicki MA. Building muscle: molecular regulation of myogenesis. Cold Spring Harb Perspect Biol. 2012 Feb 1;4(2):a008342. doi: 10.1101/cshperspect.a008342. PMID 22300977
- [Background] Brightwell CR, Latham CM, Thomas NT, Keeble AR, Murach KA, Fry CS. A glitch in the matrix: the pivotal role for extracellular matrix remodeling during muscle hypertrophy. Am J Physiol Cell Physiol. 2022 Sep 1;323(3):C763-C771. doi: 10.1152/ajpcell.00200.2022. Epub 2022 Jul 25. PMID 35876284
- [Background] Crespi EJ, Steckler TL, Mohankumar PS, Padmanabhan V. Prenatal exposure to excess testosterone modifies the developmental trajectory of the insulin-like growth factor system in female sheep. J Physiol. 2006 Apr 1;572(Pt 1):119-30. doi: 10.1113/jphysiol.2005.103929. Epub 2006 Feb 16. PMID 16484301
- [Background] Gharahdaghi N, Phillips BE, Szewczyk NJ, Smith K, Wilkinson DJ, Atherton PJ. Links Between Testosterone, Oestrogen, and the Growth Hormone/Insulin-Like Growth Factor Axis and Resistance Exercise Muscle Adaptations. Front Physiol. 2021 Jan 15;11:621226. doi: 10.3389/fphys.2020.621226. eCollection 2020. PMID 33519525
- [Background] Gonzalez ML, Busse NI, Waits CM, Johnson SE. Satellite cells and their regulation in livestock. J Anim Sci. 2020 May 1;98(5):skaa081. doi: 10.1093/jas/skaa081. PMID 32175577
- [Background] Lesnak JB, Fahrion A, Helton A, Rasmussen L, Andrew M, Cunard S, Huey M, Kreber A, Landon J, Siwiec T, Todd K, Frey-Law LA, Sluka KA. Resistance training protects against muscle pain through activation of androgen receptors in male and female mice. Pain. 2022 Oct 1;163(10):1879-1891. doi: 10.1097/j.pain.0000000000002638. Epub 2022 Mar 24. PMID 35353765
- [Background] Ringeval M, Wagner G, Denford J, Pare G, Kitsiou S. Fitbit-Based Interventions for Healthy Lifestyle Outcomes: Systematic Review and Meta-Analysis. J Med Internet Res. 2020 Oct 12;22(10):e23954. doi: 10.2196/23954. PMID 33044175
- [Background] Vleeming A, Albert HB, Ostgaard HC, Sturesson B, Stuge B. European guidelines for the diagnosis and treatment of pelvic girdle pain. Eur Spine J. 2008 Jun;17(6):794-819. doi: 10.1007/s00586-008-0602-4. Epub 2008 Feb 8. PMID 18259783
- [Result] Cong H, Liu H, Sun Y, Gao J, Liu J, Ma L, Stuge B, Chen L. Cross-cultural adaptation, reliability, and validity of a Chinese version of the pelvic girdle questionnaire. BMC Pregnancy Childbirth. 2021 Jun 30;21(1):470. doi: 10.1186/s12884-021-03962-8. PMID 34193061
- [Result] Davenport MH, Marchand AA, Mottola MF, Poitras VJ, Gray CE, Jaramillo Garcia A, Barrowman N, Sobierajski F, James M, Meah VL, Skow RJ, Riske L, Nuspl M, Nagpal TS, Courbalay A, Slater LG, Adamo KB, Davies GA, Barakat R, Ruchat SM. Exercise for the prevention and treatment of low back, pelvic girdle and lumbopelvic pain during pregnancy: a systematic review and meta-analysis. Br J Sports Med. 2019 Jan;53(2):90-98. doi: 10.1136/bjsports-2018-099400. Epub 2018 Oct 18. PMID 30337344
- [Result] Dietz HP. Ultrasound imaging of maternal birth trauma. Int Urogynecol J. 2021 Jul;32(7):1953-1962. doi: 10.1007/s00192-020-04669-8. Epub 2021 Feb 17. PMID 33595672
- [Result] Dietz HP, Shek KL. Tomographic ultrasound imaging of the pelvic floor: which levels matter most? Ultrasound Obstet Gynecol. 2009 Jun;33(6):698-703. doi: 10.1002/uog.6403. PMID 19434620
- [Result] Fagevik Olsen M, Elden H, Gutke A. Evaluation of self-administered tests for pelvic girdle pain in pregnancy. BMC Musculoskelet Disord. 2014 Apr 27;15:138. doi: 10.1186/1471-2474-15-138. PMID 24767628
- [Result] Fagevik Olsen M, Kornung P, Kallin S, Elden H, Kjellby Wendt G, Gutke A. Validation of self-administered tests for screening for chronic pregnancy-related pelvic girdle pain. BMC Musculoskelet Disord. 2021 Mar 1;22(1):237. doi: 10.1186/s12891-021-04103-0. PMID 33648489
- [Result] Ferreira CW, Alburquerque-Sendi N F. Effectiveness of physical therapy for pregnancy-related low back and/or pelvic pain after delivery: a systematic review. Physiother Theory Pract. 2013 Aug;29(6):419-31. doi: 10.3109/09593985.2012.748114. Epub 2012 Dec 17. PMID 23244038
- [Result] Marin-Jimenez N, Acosta-Manzano P, Borges-Cosic M, Baena-Garcia L, Coll-Risco I, Romero-Gallardo L, Aparicio VA. Association of self-reported physical fitness with pain during pregnancy: The GESTAFIT Project. Scand J Med Sci Sports. 2019 Jul;29(7):1022-1030. doi: 10.1111/sms.13426. Epub 2019 Apr 29. PMID 30933387
- [Result] O'Connor PJ, Poudevigne MS, Cress ME, Motl RW, Clapp JF 3rd. Safety and efficacy of supervised strength training adopted in pregnancy. J Phys Act Health. 2011 Mar;8(3):309-20. doi: 10.1123/jpah.8.3.309. PMID 21487130
- [Result] Perales M, Santos-Lozano A, Ruiz JR, Lucia A, Barakat R. Benefits of aerobic or resistance training during pregnancy on maternal health and perinatal outcomes: A systematic review. Early Hum Dev. 2016 Mar;94:43-8. doi: 10.1016/j.earlhumdev.2016.01.004. Epub 2016 Feb 3. PMID 26850782
- [Result] Petrov Fieril K, Glantz A, Fagevik Olsen M. The efficacy of moderate-to-vigorous resistance exercise during pregnancy: a randomized controlled trial. Acta Obstet Gynecol Scand. 2015 Jan;94(1):35-42. doi: 10.1111/aogs.12525. Epub 2014 Nov 13. PMID 25287282
- [Result] Sklempe Kokic I, Ivanisevic M, Uremovic M, Kokic T, Pisot R, Simunic B. Effect of therapeutic exercises on pregnancy-related low back pain and pelvic girdle pain: Secondary analysis of a randomized controlled trial. J Rehabil Med. 2017 Mar 6;49(3):251-257. doi: 10.2340/16501977-2196. PMID 28233012
- [Result] Stuge B, Jenssen HK, Grotle M. The Pelvic Girdle Questionnaire: Responsiveness and Minimal Important Change in Women With Pregnancy-Related Pelvic Girdle Pain, Low Back Pain, or Both. Phys Ther. 2017 Nov 1;97(11):1103-1113. doi: 10.1093/ptj/pzx078. PMID 29077966
- [Result] Welch N, Moran K, Antony J, Richter C, Marshall B, Coyle J, Falvey E, Franklyn-Miller A. The effects of a free-weight-based resistance training intervention on pain, squat biomechanics and MRI-defined lumbar fat infiltration and functional cross-sectional area in those with chronic low back. BMJ Open Sport Exerc Med. 2015 Nov 9;1(1):e000050. doi: 10.1136/bmjsem-2015-000050. eCollection 2015. PMID 27900136
- [Result] Wu WH, Meijer OG, Uegaki K, Mens JM, van Dieen JH, Wuisman PI, Ostgaard HC. Pregnancy-related pelvic girdle pain (PPP), I: Terminology, clinical presentation, and prevalence. Eur Spine J. 2004 Nov;13(7):575-89. doi: 10.1007/s00586-003-0615-y. Epub 2004 Aug 27. PMID 15338362